CLINICAL TRIAL: NCT02492074
Title: Gene-Environment-Interaction: Influence of the COMT Genotype on the Effects of Different Cannabinoids on the Endocannabinoid System and Brain Function
Brief Title: Gene-Environment-Interaction: Influence of the COMT Genotype on the Effects of Different Cannabinoids - a PET Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No documents were ever submitted to the Ethics Committee or the competent authority because it was not possible to establish the planned PET measurements in Germany. Therefore, the study never started.
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GEI-TCP I
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers; Modeling Psychosis
Keywords: delta-9-tetrahydrocannabinol; cannabidiol; COMT
MeSH Terms: interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- THC (Experimental): Subjects receive 20 mg delta-9-tetrahydrocannabinol (2 capsules containing 10 mg each) and corresponding cannabidiol placebo capsules.
  Interventions: Drug: Delta-9-tetrahydrocannabinol; Drug: Placebo
- CBD (Experimental): Subjects receive 800 mg cannabidiol (4 capsules containing 200 mg each) and corresponding delta-9-tetrahydrocannabinol placebo capsules.
  Interventions: Drug: Cannabidiol; Drug: Placebo
- CBD+THC (Experimental): Subjects receive 800 mg cannabidiol (4 capsules containing 200 mg each) and 20 mg delta-9-tetrahydrocannabinol (2 capsules containing 10 mg each)
  Interventions: Drug: Delta-9-tetrahydrocannabinol; Drug: Cannabidiol
- Placebo (Placebo Comparator): Subjects receive corresponding delta-9-tetrahydrocannabinol and cannabidiol placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Delta-9-tetrahydrocannabinol — oral administration of delta-9-tetrahydrocannabinol
  Other Names: Dronabinol
  Arms: CBD+THC; THC
Drug: Cannabidiol — oral administration of cannabidiol
  Arms: CBD; CBD+THC
Drug: Placebo — oral administration of placebo
  Arms: CBD; Placebo; THC

SUMMARY:
The study evaluates the gene-environment interaction of the COMT-genotype on the effects of the phytocannabinoids delta-9-tetrahydrocannabinol, cannabidiol or a combination of both on induction of psychotic symptoms, endocannabinoid levels in human body fluids, neuronal processing, and neural oscillations. In addition the effects of the phytocannabinoids on lipid levels in serum and cerebrospinal fluid, cognition, neuronal processing assessed by fMRI as well as D2-receptor availability assessed by [18F] desmethoxyfallypride.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given by the subject
* Healthy young man (age between 18 and 45) insightful to the study (WST> 95)
* Right handedness
* At least one time consumption of Cannabis but less than 10 times/ per lifetime, no consumption of other psychotropic agents (despite coffee or nicotine), no alcohol abuse
* Negative drug-screening at the time of screening
* Body Mass Index between 18 and 30

Exclusion Criteria:

* Lack of accountability
* Participation in other interventional trials
* Severe medical or neurological illness, especially cardiovascular, renal, advanced respiratory, hematological or endocrinological failures or infectious diseases (acute hepatitis A, B or C or HIV) assessed at the time of the screening by the subject's history, clinical examination and laboratory testing, at the discretion of the investigator
* Any known psychiatric illness in the participant's history
* Known family history concerning psychiatric disorders
* Cannabis consumption within the last six months
* Consumption of any illegal drugs (except cannabis in history, see above)
* Intake of interfering medication, at the discretion of the investigator
* High intracranial pressure
* Any disorders in stereoscopic vision (measured by the TNO-Test, Lamerics, Utrecht) or hearing deficits
* Contraindications due to the Investigators Brochure Contraindication for Magnetic Resonance Imaging (e.g. cardiac pacemaker, claustrophobia, attached brace, in body metal, tattoos) or lumbar puncture (e.g. local or systemic infection, disturbance of blood coagulation, medication with anticoagulants like Phenprocoumon) or contradiction for the PET-CT method and the radiopharmaceutical

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (total score, PANSS T) from baseline to post drug intake of both on induction of psychotic symptoms, endocannabinoid levels in human body fluids, neuronal processing, and D2-receptor availability | up to 6 hours

SECONDARY OUTCOMES:
Change in PANSS subscores and clusters (baseline to post drug intake) | up to 4 hours
Change in Digit Symbol Coding | up to 6 hours
Change in Letter-Number-Sequencing | up to 6 hours
Change in emotional state (EWL, "Eigenschaftswörterliste") | up to 6 hours
Change in attentional state (d2-test of attention d2-R) | up to 6 hours
Change in imagination (Bett's Questionaire upon Mental Imagery) | up to 6 hours
Change in binocular depth inversion illusion (BDII) | up to 6 hours
Change in Wisconsin Card Sorting Test Performance | up to 6 hours
Assessment of hallucinogenic states scale (APZ) (post drug intake) | 1 day
  questionaire
Safety and tolerability assessments including (S)AEs, physical examination, vital signs (including heart rate and systolic and diastolic blood pressure in both supine and standing positions), and detailed laboratory assessments | 1 day
Metabolic markers post drug intake (blood) | up to 4 hours
Metabolic markers post drug intake (cerebrospinal fluid) | up to 4 hours
D2-receptor availability post drug intake | up to 5 hours

OTHER OUTCOMES:
Assessment of biomarker profiles in serum and cerebrospinal fluid of subjects | 1 day
  Comparison of biomarker profiles in serum and cerebrospinal fluid after different treatments

CONTACTS AND LOCATIONS:
Overall Officials: F. Markus Leweke, MD, Principal Investigator — Central Institute of Mental Health
Locations (1):
- Central Institute of Mental Health, Mannheim, Baden-Wurttemberg, Germany